CLINICAL TRIAL: NCT01318460
Title: Prophylactic Administration of Levosimendan in Patients With Impaired Left Ventricular Function Undergoing Coronary Surgery
Brief Title: Prophylactic Administration of Levosimendan in Patients Undergoing Coronary Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AHEPA University Hospital (Other)
Collaborators: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Principal Investigator, Kyriakos Anastasiadis, Head of Cardiothoracic Department, AHEPA University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AHEPA_CTS-03
Record Dates: First submitted 2011-03-17; First posted 2011-03-18 (Estimated); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Coronary Artery Disease
Keywords: coronary artery disease; levosimendan; coronary artery bypass grafting; cardiac surgery
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Levosimendan (Active Comparator): Patients treated with prophylactic administration of levosimendan
  Interventions: Drug: Levosimendan infusion
- Placebo group (Placebo Comparator): Patients managed with placebo administration
  Interventions: Drug: Placebo infusion

INTERVENTIONS:
Drug: Levosimendan infusion — Prophylactic 24h infusion of levosimendan at a dose of 0.1 mg/kg/min
  Arms: Levosimendan
Drug: Placebo infusion — Twenty-four hour administration of placebo
  Arms: Placebo group

SUMMARY:
The present pilot study aims to investigate the effectiveness of the preoperative infusion of levosimendan in patients with impaired left ventricular function undergoing coronary artery bypass grafting.

DETAILED DESCRIPTION:
Myocardial revascularization in patients with impaired left ventricular function remains a serious problem in cardiac surgery. Despite the recent developments with the use of new surgical techniques (mini-extracorporeal circulation, off pump surgery) the perioperative morbidity and mortality are relatively high. Therapeutic solutions with the use of inotropic drugs, as adrenergic agonists and phosphodiesterase inhibitors, have offered important improvement to the hemodynamic status of these patients, but they have not considerably decreased mortality. These drugs owe their positive inotropic action to the increase of intracellular calcium and thereafter they improve the myocardial function.

Levosimendan (SIMDAX) is a new calcium sensitizer which increases the myocardial contractility without particular promotion of the intracellular calcium accumulation. Contemporary experimental and clinical data demonstrated the effectiveness of this drug in the reduction of surgical mortality to the patients with low left ventricular ejection fraction (LVEF) who undergo coronary artery bypass grafting (CABG).

This is an original prospective randomized controlled study focused on the preoperative use of this drug in patients with impaired left ventricular function which is associated with a high operative risk (i.e. EuroSCORE). Perioperative myocardial stunning is particularly evident in this cohort of patients. Prophylactic administration of levosimendan the day before the operation could be translated in improved myocardial performance intraoperatively and during the early postoperative period.

ELIGIBILITY:
Inclusion Criteria:

* coronary artery disease which warrants myocardial revascularization with coronary artery bypass grafting according to current guidelines
* age < 79 years old
* left ventricular ejection fraction <= 40%
* informed patient's consent

Exclusion Criteria:

* age < 18 years old
* emergency surgery
* medical history of acute myocardial infarction with ST elevation (STEMI) less than 14 days old
* any severe comorbidity which increases the perioperative risk (i.e. neoplasia, rheumatoid arthritis, chronic obstructive pulmonary disease)
* need for valvular replacement surgery
* redo surgery
* serum creatinine > 2 mg/dl
* history of malignant cardiac arrhythmias

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2011-03; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Left ventricular function | Seventh postoperative day
  Left ventricular function as assessed by transthoracic or transesophageal echocardiography on the seventh postoperative day

SECONDARY OUTCOMES:
Perioperative mortality | 30 days postoperatively
Need for intraaortic balloon pump | 1st-7th postoperative day
Inotropic support | 1st-7th postoperative day
  Need for high inotropic support
Total ICU stay | 1st-7th postoperative day
Total length of hospital stay | 1st-7th postoperative day
Time on mechanical ventilation | 1st-7th postoperative day
Major adverse cardiovascular events | 1st-7th postoperative day
  Perioperative myocardial infarction, stroke, need for revascularization)
Morbidity | 1st-7th postoperative day

CONTACTS AND LOCATIONS:
Overall Officials: Kyriakos Anastasiadis, MD, FETCS, Principal Investigator — AHEPA University Hospital; Christos Papakonstantinou, MD, Study Chair — AHEPA University Hospital
Locations (1):
- Department of Cardiothoracic Surgery, AHEPA University Hospital, Thessaloniki, Greece

REFERENCES:
- [Background] De Hert SG, Lorsomradee S, Cromheecke S, Van der Linden PJ. The effects of levosimendan in cardiac surgery patients with poor left ventricular function. Anesth Analg. 2007 Apr;104(4):766-73. doi: 10.1213/01.ane.0000256863.92050.d3. PMID 17377079
- [Background] Tasouli A, Papadopoulos K, Antoniou T, Kriaras I, Stavridis G, Degiannis D, Geroulanos S. Efficacy and safety of perioperative infusion of levosimendan in patients with compromised cardiac function undergoing open-heart surgery: importance of early use. Eur J Cardiothorac Surg. 2007 Oct;32(4):629-33. doi: 10.1016/j.ejcts.2007.07.010. Epub 2007 Aug 15. PMID 17702589
- [Background] Kolseth SM, Nordhaug DO, Stenseth R, Sellevold O, Kirkeby-Garstad I, Wahba A. Prophylactic treatment with levosimendan: a retrospective matched-control study of patients with reduced left ventricular function. Eur J Cardiothorac Surg. 2009 Dec;36(6):1024-30. doi: 10.1016/j.ejcts.2009.05.001. Epub 2009 Jul 9. PMID 19592266